CLINICAL TRIAL: NCT06532851
Title: The Efficacy of Progressive Resistance Exercises Versus Aerobic Exercises on Cartilage Morphology and Physical Function in Patients With Degenerative Meniscus Tear: A Randomized Controlled Trial
Brief Title: The Effect of Therapeutic Exercise on Cartilage Morphology and Physical Function for Individuals at High Risk of Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230630
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Meniscus Tear
Keywords: Degenerative Meniscus Tear; MRI T2 Mapping; Progressive Resistance Exercise; Aerobic Exercise; Knee Pain; Cartilage Morphology; Exercise Therapy; Early Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy; Resistance Training; Exercise

STUDY DESIGN:
Intervention Model Description: In this model, participants are assigned to one of the three groups (PRE, aerobic exercise, control) and remain in that group for the duration of the study. Each group receives a different intervention, allowing for direct comparisons between the interventions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this study, the outcomes assessor and the investigators will be blinded to the group allocation. The outcomes assessor will be unaware of the participants' group assignments to minimize the potential bias in evaluating outcomes. Similarly, the treatment assignment will only be displayed to the principal investigator once it has been determined that the subject meets all eligibility criteria, thus preserving concealed allocation of the randomization assignment from the study investigators and the individuals responsible for subject recruitment and follow-up. To minimize bias throughout the study, individuals responsible for collecting the outcome measures will remain blinded to group assignment for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive Resistance Exercise (PRE) (Experimental): Participants will perform progressive resistance exercises focusing on strengthening the quadriceps muscles. The exercises will be adjusted based on the Daily Adjustable Progressive Resistance Exercise (DAPRE) technique.
  Interventions: Other: Progressive Resistance Exercise (PRE)
- Aerobic Exercise (Experimental): Participants will engage in aerobic exercise sessions using a stationary bike, aimed at improving cardiovascular fitness and knee joint mobility.
  Interventions: Other: Aerobic Exercise
- Control (Active Comparator): Participants will receive standard of care, including general strength and balance exercises as per current clinical guidelines.
  Interventions: Other: Control

INTERVENTIONS:
Other: Progressive Resistance Exercise (PRE) — A structured exercise regimen focusing on increasing muscular strength and endurance through progressive resistance.
  Other Names: Exercise Therapy; Resistance Training
  Arms: Progressive Resistance Exercise (PRE)
Other: Aerobic Exercise — An exercise program focusing on cardiovascular conditioning using a stationary bike.
  Other Names: Exercise Therapy; Aerobic Training
  Arms: Aerobic Exercise
Other: Control — A set of general strength and balance exercises that do not target the specific therapeutic goals of the other interventions.
  Other Names: Comparator
  Arms: Control

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy of progressive resistance exercises (PRE) versus aerobic exercises on cartilage morphology and physical function in patients with degenerative meniscus tears. 54 participants, aged 35-55, will be randomly assigned to one of three groups: PRE, aerobic exercise, or control (standard of care physical and medical therapy). The study will utilize MRI T2 mapping to assess changes in cartilage composition and patient-reported and performance-based measures to evaluate clinical outcomes. This pilot study will also determine the feasibility and issues related to recruitment and retention for a larger trial.

DETAILED DESCRIPTION:
Background: Degenerative meniscus tears are common in individuals over 35 and are associated with early stages of knee osteoarthritis (OA) (1,2). Metabolic and microstructural changes within the cartilage occur before surface breakdown, which can now be detected using advanced MRI techniques such as T2 mapping. Exercise therapy, specifically progressive resistance and aerobic exercises, has shown benefits for knee OA patients, but its effects on early cartilage degeneration are poorly understood.

Objective: The primary objective of this study is to determine the efficacy of PRE and aerobic exercises on the metabolic function and microstructure of cartilage in individuals with degenerative meniscus tears but without radiographic evidence of knee OA. Secondary objectives include evaluating the impact of these exercises on clinical outcomes, such as pain, disability, and physical function, and assessing the feasibility of recruitment and retention for a larger trial.

Methods: The study will enroll 54 participants, who will be randomized into three groups: PRE, aerobic exercise, and control. Each group will undergo a 3-month supervised exercise program. MRI scans will be used to measure changes in cartilage composition, while clinical outcomes will be assessed using patient-reported and performance-based measures.

Intervention Groups:

Group 1 (PRE): Participants will perform progressive resistance exercises focusing on strengthening the quadriceps. The exercises will be adjusted based on the Daily Adjustable Progressive Resistance Exercise (DAPRE) technique.

Group 2 (Aerobic Exercise): Participants will engage in aerobic exercise sessions using a stationary bike, aimed at improving cardiovascular fitness and knee joint mobility.

Group 3 (Control): Participants will receive standard of care, including general strength and balance exercises as per current clinical guidelines.

Assessments:

MRI Imaging: Advanced MRI techniques (T2 mapping) will be used at baseline and after 3 months to assess changes in cartilage composition.

Clinical Outcomes: Patient-reported outcomes will include the Knee Injury and Osteoarthritis Outcome Score (KOOS) and the International Knee Documentation Committee (IKDC) score. Performance-based outcomes will include the single-leg squat, single-leg hop test, sit-to-stand on a one-foot test, step-up test, and Bruce treadmill test.

Inclusion Criteria:

Adults aged 35-55 years Symptomatic degenerative medial meniscus tears. No radiographic evidence of knee OA (Kellgren-Lawrence grade 0-1). Ability to provide informed consent. Willingness to participate in the exercise intervention.

Exclusion Criteria:

Existing diagnosis of knee OA (Kellgren-Lawrence grade 2 or higher). Repairable meniscus injuries or prior meniscus repair. Previous knee surgery or significant knee injury within the past 6 months. Presence of inflammatory arthritis or other significant comorbidities. Contraindications to MRI or inability to participate in exercise programs.

Study Outcomes:

Primary Outcomes: Changes in T2 relaxation times in the cartilage, indicating alterations in cartilage composition and health.

Secondary Outcomes: Improvements in clinical outcomes, including pain, disability, and physical function as measured by KOOS, IKDC, and performance-based tests.

Feasibility Metrics: Recruitment rates, adherence to the exercise program, and retention rates over the study period.

Analysis: A mixed ANOVA will be used to compare changes in outcomes between groups, with adjustments for multiple comparisons. Baseline characteristics will be compared using t-tests and chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

1. Are between 35 and 55 years of age.
2. Have a symptomatic degenerative medial meniscus tear as evidenced by:

   * Presence of medial knee pain.
   * Medial joint line tenderness.
   * Pain and limited motion when attempting to perform a full squat and
   * Increased intra-meniscal signal on at least 2 consecutive MRI slices and
3. Have clearance from their personal physician to participate in an exercise program.

Exclusion Criteria:

1. Radiographic evidence of OA (K-L grade 2 or above).
2. A repairable meniscus injury (longitudinal tear in the outer 1/3 of the meniscus).
3. A meniscus injury that requires meniscectomy (locked knee).
4. Prior or current ligament injury or surgery of the involved knee.
5. Prior or current injury or surgery to contra-lateral knee.
6. Pathological ligamentous laxity upon examination of the knee
7. An inflammatory arthritic condition or
8. Any injury or condition involving the lower extremities that affects their ability to walk.

Because participation in this study requires undergoing MRI, subjects will be excluded if they:

1. If female, pregnant at the time of enrollment.
2. Had prior surgery for an aneurysm; any medical illness that may interfere with the patient's general fitness or exercise capability.
3. Had any contraindication with MRI.
4. Had surgery within the past two months.
5. Have a cardiac pacemaker.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Short echo T2* | Baseline, 3-month, 12-month, and 5 years follow-ups.
  Short echo time T2* imaging is used to diagnose early cartilage degeneration. T2* measures the rate at which the MRI signal decays, particularly focusing on short-T2 signals (less than 10 milliseconds) which decay rapidly (3-6).

SECONDARY OUTCOMES:
Single leg hop test for a distance | Baseline, immediately post-intervention, 3-month, 6-month, 12-month, and 5 years follow-ups.
  The Single Leg Hop Test for distance is one of four assessments used to evaluate athletes' horizontal movement capabilities. These tests, collectively known as the 4 Single Leg Hop Tests, were established by Noyes et al (7). They include the Triple Hop for distance, the Single Leg Hop Test for distance, the 6-meter hop for time, and the Crossover Hop for distance.
  In the Single Leg Hop Test for distance, participants stand on one leg with their toes aligned along a designated landmark line. They then execute a forward hop, landing eccentrically while maintaining balance on the tested leg. The examiner measures the distance from the initial landmark line to the point where the participant's heel contacts the ground (8).
  This test is valuable for assessing lower extremity strength, power, and balance. It has been shown to be a reliable and valid measure for evaluating aspects of lower extremity function (9-10).
Single Leg Squat Test | Baseline, immediately post-intervention, 3-month, 6-month, 12-month, and 5 years follow-ups.
  The Single Leg Squat Test is a functional movement assessment used to evaluate lower extremity strength, neuromuscular control, and stability. Beyond its focus on lower limb function, it also helps identify core muscle strength and provides insights into an individual's capabilities in cutting, running, and landing (11). The SLST assesses the ability to alternate between concentric and eccentric contractions of the knee and hip muscles (12).
  In the test, the patient stands on one leg with their foot aligned with a straight line. The examiner assists with balance and ensures proper form. The patient then performs knee bends until the line along their toes is no longer visible, within a 30-degree range of knee flexion. Each patient has 30 seconds to complete as many repetitions as possible, with the maximum number recorded (13-16). The physiotherapist monitors and adjusts the test to maintain accuracy and consistency.
The Timed Stair Climbing Test (SCT) | Baseline, immediately post-intervention, 3-month, 6-month, 12-month, and 5 years follow-ups.
  The Timed Stair Climbing Test (SCT) is a functional performance assessment designed to evaluate lower extremity strength, endurance, and functional mobility. Participants will ascend and descend a 12-step staircase, with each step measuring 18 cm in height and 28 cm in depth. The objective is to complete the test as quickly as possible while ensuring a sense of safety and comfort. While the use of one handrail is optional, participants are encouraged to refrain from using it (17).
The Single Leg Chair Rise (SLCR) test | Baseline, immediately post-intervention, 3-month, 6-month, 12-month, and 5 years follow-ups.
  The Single Leg Chair Rise (SLCR) test evaluates quadriceps strength and can also help diagnose mid-lumbar nerve root impingement and radiculopathy (18,19). It has a sensitivity of 0.48, a specificity of 0.90, a positive likelihood ratio of 4.60, and a negative likelihood ratio of 0.58 (19).
  The protocol uses a 45.7 cm chair. Participants, dressed and shod, sit with arms crossed, the tested leg flexed at 90 degrees, and the other leg extended without touching the ground. They rise to full knee extension and then return to the seated position to complete one repetition. The test includes two assessments: one measuring endurance with as many repetitions as possible in 30 seconds, and another measuring power by completing five repetitions as quickly as possible. Each test is performed twice, with the best score recorded (20).
Maximal voluntary isometric contraction test | Baseline, immediately post-intervention, 3-month, 6-month, 12-month, and 5 years follow-ups.
  To assess quadriceps muscle strength, the maximum voluntary isometric torque test will be performed using an isokinetic dynamometer (Biodex System 3 Pro). The procedure involves the participant seated with their ankle positioned in line with the dynamometer's axis at 60 degrees of knee flexion, secured by waist, thigh, and chest straps (21).
  Before testing, participants will familiarize themselves with the process by performing isometric contractions at 50%, 75%, and 100% of their maximal effort. During the actual test, they will exert maximal force against the dynamometer's fixed arm for knee extension. Each participant will complete three trials with a two-minute rest between them, aiming to match or exceed a target torque displayed on a screen. The target torque will be adjusted based on their performance in previous trials. The maximum quadriceps muscle strength will be calculated using the recorded data (21).
The Modified Bruce Treadmill Testing Protocol | Baseline, immediately post-intervention, 3-month, 6-month, 12-month, and 5 years follow-ups.
  The modified Bruce Test is designed for sedentary and elderly patients to estimate maximal oxygen consumption (VO2max) and assess aerobic endurance. Unlike the standard Bruce Test, which includes seven stages of increasing speed and incline on a treadmill, the modified version starts with a lower workload. It begins at 1.7 km/hr with a 0% incline and progresses to a 5% incline in the second stage, before resembling the first stage of the standard test. This modified approach includes "Stage Zero" and "1/2" to indicate the initial zero incline and a slight incline in the following stage, making it more suitable for less fit individuals (22,23).
  VO2max measures the maximum amount of oxygen a person uses during intense exercise. It is calculated based on the duration of exercise using different formulas for men and women, without needing to measure inhaled and exhaled air directly (22,23):
  Women: VO2max (ml/kg/min) = 4.38 × T - 3.9 Men: VO2max (ml/kg/min) = 2.94 × T + 7.65
International Knee Documentation Committee Subjective Knee Form (IKDC) | Baseline, immediately post-intervention, 3-month, 6-month, 12-month, and 5 years follow-ups.
  The International Knee Documentation Committee Subjective Knee Form (IKDC) was developed in 2001 through a collaboration between the European Society for Sports Traumatology, Knee Surgery, and Arthroscopy, and the American Orthopaedic Society for Sports Medicine (AOSSM). This form is a widely used patient-reported outcome measure that assesses subjective aspects of a patient's health related to knee conditions. It includes domains such as symptoms, functional limitations, and sports activities. The IKDC has been translated into numerous languages, including Arabic for this study. It comprises ten questions, with one evaluating the impact of the knee on daily activities and nine focusing on performance. Scores range from 0 to 100, with higher scores indicating better health status (24).
The Knee injury and Osteoarthritis Outcomes Score (KOOS) | Baseline, immediately post-intervention, 3-month, 6-month, 12-month, and 5 years follow-ups.
  The Knee Injury and Osteoarthritis Outcomes Score (KOOS) is a patient-reported outcome measure designed to assess the impact of knee injury or osteoarthritis on an individual's quality of life (25,26). It includes subscales for pain, symptoms, activities of daily living (ADL), quality of life, and recreational activities (25,26). Studies have shown that KOOS has superior psychometric characteristics compared to other measures. It has been translated into 40 languages, including an Arabic version for use in Saudi Arabia, which will be utilized in our study (27,28). KOOS comprises 42 items across five subscales: nine for pain, seven for symptoms, seventeen for ADL, five for sports and recreation function, and four for knee-related quality of life. Each item is scored from 0 to 4, with higher scores indicating better health status (29).

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - King Abdullah University Hospital, Ar Ramtha
  - Jordan University of Science and Technology, Irbid

REFERENCES:
- See also: (1) Englund M, Roos EM, Roos HP, Lohmander LS. Patient-relevant outcomes fourteen years after meniscectomy: influence of type of meniscal tear and size of resection. Rheumatology. 2001 Jun;40(6):631-9. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (2) Wolf BR, Gulbrandsen TR. Degenerative Meniscus Tear in Older Athletes. Clin Sports Med. 2020 Jan;39(1):197-209. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (3) Carlier PG, Bertoldi D, Baligand C, Wary C, Fromes Y. Muscle blood flow and oxygenation measured by NMR imaging and spectroscopy. NMR Biomed. 2006 Nov;19(7):954-67. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (4) Gatehouse PD, Bydder GM. Magnetic Resonance Imaging of Short T2 Components in Tissue. Clin Radiol. 2003 Jan;58(1):1-19. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (5) Gatehouse PD, Thomas RW, Robson MD, Hamilton G, Herlihy AH, Bydder GM. Magnetic resonance imaging of the knee with ultrashort TE pulse sequences. Magn Reson Imaging. 2004 Oct;22(8):1061-7. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (6) Qian Y, Boada FE. Acquisition-weighted stack of spirals for fast high-resolution three-dimensional ultra-short echo time MR imaging. Magn Reson Med. 2008 Jul;60(1):135-45. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (7) NOYES, F.R., S.D. BARBER, AND R.E. MANGINE. Abnormal lower limb symmetry determined by functional hop tests after anterior cruciate ligament rupture. Am. J. Sports Med. 19:513-518. 1991. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (8) Ross MD, Langford B, Whelan PJ. Test-retest reliability of 4 single-leg horizontal hop tests. J Strength Cond Res. 2002 Nov;16(4):617-22. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (9) BOLGLA, L.A., AND D.R. KESKULA. Reliability of lower extremity functional performance tests. J. Orthop. Sports Phys. Ther. 26:138- 142. 1997. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (10) BOOHER, L.D., K.M. HENCH, T.W. WORRELL, AND J. STIKELEATHER. Reliability of three single-leg hop tests. J. Sport Rehab. 2:165- 170. 1993. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (11) Ugalde V, Brockman C, Bailowitz Z, Pollard CD, Single Limb Squat Test and its Relationship to Dynamic Knee Valgus and Injury Risk Screening, PM&R (2014), doi: 10.1016/ j.pmrj.2014.08.361. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (12) Ageberg E, Bennell KL, Hunt MA, Simic M, Roos EM, Creaby MW. Validity and inter-rater reliability of medio-lateral knee motion observed during a single-limb mini squat. BMC Musculoskelet Disord. 2010 Nov 16;11:265. doi: 10.1186/1471-2474-11-265. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (13) Roos EM, Bremander AB, Englund M, Lohmander LS. Change in self-reported outcomes and objective physical function over 7 years in middle-aged subjects with or at high risk of knee osteoarthritis. Ann Rheum Dis. 2008 Apr;67(4):505-10. doi: 10.1136/ — http://pubmed.ncbi.nlm.nih.gov/
- See also: (14) Bremander AB, Dahl LL, Roos EM. Validity and reliability of functional performance tests in meniscectomized patients with or without knee osteoarthritis. Scand J Med Sci Sports. 2007 Apr;17(2):120-7. doi: 10.1111/j.1600-0838.2006.00544.x. PMID: 1 — http://pubmed.ncbi.nlm.nih.gov/
- See also: (15) Roos EM, Ostenberg A, Roos H, Ekdahl C, Lohmander LS. Long-term outcome of meniscectomy: symptoms, function, and performance tests in patients with or without radiographic osteoarthritis compared to matched controls. Osteoarthritis Cartilage 2001 — http://pubmed.ncbi.nlm.nih.gov/
- See also: (16) Stensrud S, Risberg MA, Roos EM. Knee function and knee muscle strength in middle-aged patients with degenerative meniscal tears eligible for arthroscopic partial meniscectomy. Br J Sports Med. 2014 May;48(9):784-8. doi: 10.1136/bjsports-2012-091 — http://pubmed.ncbi.nlm.nih.gov/
- See also: (17) Mizner RL, Petterson SC, Stevens JE, Axe MJ, Snyder-Mackler L. Preoperative quadriceps strength predicts functional ability one year after total knee arthroplasty. J Rheumatol. 2005 Aug;32(8):1533-9. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (18) Rainville J, Jouve C, Finno M, Limke J. Comparison of four tests of quadriceps strength in l3 or l4 radiculopathies. Spine. 2003;28(21):2466-2471. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (19) Suri P, Rainville J, Katz JN, et al. The accuracy of the physical examination for the diagnosis of midlumbar and low lumbar nerve root impingement. Spine. 2011;36(1):63-73. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (20) Waldhelm A, Gubler C, Sullivan K, Witte C, Buchheister D, Bartz-Broussard J. INTER-RATER AND TEST-RETEST RELIABILITY OF TWO NEW SINGLE LEG SIT-TO-STAND TESTS. Int J Sports Phys Ther. 2020 May;15(3):388-94. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (21) Fitzgerald GK, Piva SR, Irrgang JJ. A modified neuromuscular electrical stimulation protocol for quadriceps strength training following anterior cruciate ligament reconstruction. J Orthop Sports Phys Ther. 2003 Sep;33(9):492-501. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (22) Bruce RA. Methods of exercise testing. Step test, bicycle, treadmill, isometrics. Am J Cardiol. 1974 May 20;33(6):715-20. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (23) McInnis KJ, Balady GJ. Comparison of submaximal exercise responses using the Bruce vs modified Bruce protocols. Med Sci Sports Exerc. 1994 Jan;26(1):103-7. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (24) Almalki H, Herrington L, Jones R. Arabic version of the International Knee Documentation Committee Subjective Knee Form (IKDC): Translation and validation. J Back Musculoskelet Rehabil. 2022;35(3):659-65. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (25) Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD (1998) Knee Injury and Osteoarthritis Outcome Score (KOOS)- development of a self-administered outcome measure. J Orthop Sports Phys Ther 28:88-96. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (26) Roos EM, Lohmander LS (2003) The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes 1:64-68. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (27) Garratt AM, Brealey S, Gillespie WJ (2004) Patient-assessed health instruments for the knee: a structured review. Rheumatology 43:1414-1423. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (28) Bekkers JE, de Windt TS, Raijmakers NJ, Dhert WJ, Saris DB (2009) Validation of the Knee Injury and Osteoarthritis Outcome Score (KOOS) for the treatment of focal cartilage lesions. Osteoarthr Cartil 17:1434-1439. — http://pubmed.ncbi.nlm.nih.gov/
- See also: (29) Alfadhel SA, Vennu V, Alnahdi AH, Omar MT, Alasmari SH, AlJafri Z, et al. Cross-cultural adaptation and validation of the Saudi Arabic version of the Knee Injury and Osteoarthritis Outcome Score (KOOS). Rheumatol Int. 2018 Aug 7;38(8):1547-55. — http://pubmed.ncbi.nlm.nih.gov/